CLINICAL TRIAL: NCT06753942
Title: ANTI-SARS-CoV-2 SEROCONVERSIO IN IMMUNE-MEDIATED KIDNEY DISEASES
Acronym: SIERO-MRI
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SIERO-MRI
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Immune-mediated Diseases; Glomerulonephritis
Keywords: immune-mediated kidney disease; seroconversion; antiSARS Cov-2 vaccination
MeSH Terms: conditions — Glomerulonephritis; HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicentric, observational, retrospective study. The primary endpoint of the study is to investigate the humoral immunological response to SARS-Cov-2 vaccination in this population, looking for clinical features predisposing to seroconversion failure.

Secondary endpoints are

* to investigate the appearance of symptomatic SARS-CoV-2 infection, despite vaccination, looking for any clinical features predisposing to infection,
* to identify the protective cut-off of antibody titer against SARS-CoV-2 infection.

Each study participating center will select all vaccinated patients with immune-mediated renal diseases for whom anti-COVID serology will be available.

DETAILED DESCRIPTION:
SARS-CoV-2 infection produces a quantifiable immune response. Post-infection immunity consists of a humoral and cell-mediated response, which appears to reduce the risk of SARS-CoV-2 re-infection for at least 6 months in the healthy population. It is reasonable to assume that SARS-COV-2 vaccination may also induce a similar response.

In immunomediated renal disease patients, it is not known what the antibody response is, what factors can potentially influence it, other than immunosuppressive therapy. This information, on the other hand, is useful not only in identifying individuals at risk of infection despite vaccination but it can help to personalize the vaccination schedule.

All patients with immune-mediated renal diseases undergoing the complete vaccination cycle (one or two doses depending on the type of vaccine used) against SARS-CoV-2, and for whom at least one dosage of anti-SARS-CoV-2 antibodies are eligible.

After obtaining signed informed consent, personal data, underlying disease, biochemical parameters (including immunoglobulin assay and lymphocyte typing, if available), present or previous comorbidities, immunosuppressive therapies, dosage of SARS-CoV-2 IgG antiSpike and/or antiRBD/Spike antibodies, the date of vaccinations and the type of vaccine performed will be extracted.

The data are all present in the patients' inpatient and/or outpatient medical records, as part of normal clinical management and completely independent of participation in the current clinical trial.

The interview with the patient will show the possible appearance of COVID-19 infection, the date of his diagnosis, confirmed by a positive molecular swab, the degree of severity and the clinical course.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 years 2. MRI diagnosis (biopsy and non-biopsy) 3. At least one complete vaccination cycle according to the indications of the NHS (consisting of two doses or a single dose depending on the type of vaccine) 4. Signing of informed consent 5. At least one dose of anti-SARS-CoV2 IgG antibodies performed after a complete vaccination course

Exclusion Criteria:

* SARS-CoV-2 infection, before or during the vaccination cycle (between I and II dose), diagnosed by molecular swab or positivity to anti-Nucleocapsid antibodies or anti-Spike IgM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with immune-mediated renal diseases undergoing the complete vaccination cycle (one or two doses depending on the type of vaccine used) against SARS-CoV-2, and for whom at least one dosage of anti-SARS-CoV-2 antibodies is available.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion for antiSARS-CoV-2 antibodies | 12 months from first vaccination
  % of MRI patients with seroconversion for antiSARS-CoV-2 antibodies and the antibody titer figure expressed as the number of SARS-CoV-2 IgG antiSpike or antiRBD/Spike antibodies.

SECONDARY OUTCOMES:
SARS Cov-2 infection despite vaccination | 12 months from first vaccination
  % of MRI patients who will develop a symptomatic SARS-CoV-2 infection will be calculated.
Antibody titer against SARS-CoV-2 infection | 12 months from first vaccination
  to identify the protective cut-off of antibody titer against SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Fausta Catapano, MD, PhD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No